CLINICAL TRIAL: NCT02370732
Title: Alcohol Related Impairment and Reinforcement After Gastric Bypass Surgery
Brief Title: Alcohol Related Impairment and Reinforcement: Pre to Post Roux en Y Gastric Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: University of Kentucky (Other); Kent State University (Other); North Dakota State University (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Research Scientist, Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AA022336
Record Dates: First submitted 2015-02-12; First posted 2015-02-25 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Bariatric Surgery Candidate
Keywords: Alcohol; Bariatric Surgery; Roux en Y Gastric bypass; Alcohol impairment; Alcohol reinforcement; Alcohol pharmacokinetics
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roux en Y Gastric Bypass (Other): Participants recruited for this protocol will be those planning to undergo Roux-en-Y Gastric Bypass (RYGB). Upon study screening completion, participants will take part in a total of 4 laboratory assessment days where a fixed dose of alcohol will be given.
  * 2 pre-surgery research appointments where participants will be given alcohol: a driving simulator day and a cognitive testing and reinforcement testing day.
  * 2 post-surgery (1 year) research appointments where you will be given alcohol: a driving simulator day and a cognitive testing and reinforcement testing day.
  Interventions: Other: Alcohol

INTERVENTIONS:
Other: Alcohol — A weight based dose of alcohol will be administered during each study day.

SUMMARY:
The proposed project will help to understand the changes in reinforcement and impairment experienced by Roux en Y bariatric surgery (RYGB) patients who consume alcohol. In this study the investigators propose to investigate RYGB patients with a prospective, longitudinal design. Investigators will examine driving impairment before and after surgery as well as study cognitive changes and reinforcement changes that may occur in RYGB patients while consuming alcohol. Finally, investigators aim to better characterize the changes that occur in the pharmacokinetics of alcohol following bariatric surgery and examine key variables which may play a role in the development in alcohol use disorders.

DETAILED DESCRIPTION:
The three major objectives of this NIH sponsored application are: 1) to characterize the severity of cognitive impairment and driving performance changes following alcohol consumption in a group of patients who have undergone Roux-en-Y Gastric Bypass (RYGB) bariatric surgery and 2) to investigate differential reinforcing properties of alcohol in patients before and after they undergo RYGB. Both of these objectives stem from observations from the investigators work and previous empirical studies suggesting that the pharmacokinetics (PK) of alcohol are substantially altered following bariatric surgery. This may lead to alterations in the time-course and severity of alcohol-related cognitive and driving impairment, as well as alter the reinforcing effects of drinking alcohol. Particularly relevant to these objectives, PK data have shown higher peak alcohol concentrations and a shorter time to achieve them in bariatric surgery patients. Therefore the third objective of this application is to better characterize the PK profile of alcohol following RYGB. Finally, investigators will explore whether changes in impairment, reinforcement, and PKs are moderated by gender, age, smoking, and alcohol use.

In this study investigators propose to prospectively investigate approximately 50-60 RYGB patients. Participants will be assessed at baseline (pre-surgery) and one year after surgery (to approximate their weight nadir) in an acute alcohol dosing laboratory paradigm.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (approximately 50% each)
2. 21 - 65 years of age
3. In evaluation for Roux-en-Y gastric bypass surgery
4. Able to tolerate alcohol dose
5. Cognitive ability to complete study protocol as assessed at screening
6. Medically stable

Exclusion Criteria:

1. History of or current alcohol use disorder (as assessed at screening)
2. Psychotic or bipolar spectrum disorder (as assessed at screening)
3. Current suicidality (as assessed at screening)
4. Concomitant medication known to significantly interact with alcohol
5. Concomitant medication known to significantly impact driving simulator performance
6. Pregnancy or intending to become pregnant prior to the end of the their participation in the study or breastfeeding
7. Positive urine drug screen
8. Unable to tolerate blood draws
9. Significant risk for developing motion sickness while using the driving simulator
10. Unable to speak English
11. Other factor that would increase participant risk in the protocol in the judgement of the investigators or physician.
12. Participated in an investigational drug study within the past 30 days
13. Is or has an immediate family member that is employeed by the Neuropsychiatric Research Institute
14. Has a pacemaker
15. Insulin dependent diabetes mellitus
16. Smoking defined as regular use of nicotine in the past 6 months
17. A presurgery weight of > 400lbs at screening appointment or as reported on telephone screen
18. Unable to provide a blood sample at the screening appointment or is assessed to have poor vein quality for IV placement as determined by the research clinical personnel.
19. Laboratory abnormalities defined as a hepatic panel greater than three times the upper limit of normal, or fasting glucose of < 60 or >120 mg/dl, or positive pregnancy test.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in Drive Safety RS-300 Research Driving Simulator Performance | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  We will be assessing participants for evidence of a change in driving impairment using the Drive Safety RS-300 Research Driving Simulator, which provides a high-quality, authentic automotive control environment based on a midsized Ford Focus passenger car. The simulation is controlled by a bank of computers running DriveSafety's Vection software, which enables real-time data collection and updating of the displays. DriveSafety's HyperDrive Authoring Suite is used to model complex driving scenarios and to precisely control the presentation of stimuli within the simulated environment.

SECONDARY OUTCOMES:
Change in Desire-for-Drug Scale | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The Desire-for-Drug Scale is a 4-item VAS measure commonly used in research on alcohol priming effects that study increases in motivation to drink after a dose of alcohol (e.g., Fillmore, 2001). The scale measures the motivation to consume alcohol (i.e., priming), assesses subjective ratings of its effect, and is viewed as an indicator of the reward a person associates with alcohol consumption. The measure of priming is assessed by an item that asks participants how much they "have a desire for alcohol".
Change in pharmacokinetics as measured via blood alcohol concentrations | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  Pharmacokinetic assessments of alcohol plasma levels and will be analyzed using model-independent (noncompartmental) methods with the use of Phoenix WinNonlin® Version 6.1 (Pharsight, Mountain View, CA).
Change in 2-Back task | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  We will be assessing cognitive impairment using the 2-Back task. This task is a complex working memory task in which a series of 15 consonants is presented visually. Participants are asked to make a yes/no response following each consonant - whether it is the same as, or different from, the consonant presented two earlier.

OTHER OUTCOMES:
Change in Structured Clinical Interview for DSM (SCID-I/P; First et al., 1995) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The SCID-I/P will provide a thorough assessment of Axis I psychopathology in order to examine the impact of co-occurring psychiatric disorders on the parameters of interest.
Change in Addiction Severity Index (ASI) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The ASI will be used to carefully examine alcohol and drug abuse frequency and severity
Change in Alcohol Use Disorders Identification Test (AUDIT; Barbor, et al., 2001) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The AUDIT is a ten-item measure developed by the World Health Organization to assess alcohol use and alcohol-related consequences.
Change in Michigan Alcohol Screening Test (MAST; Selzer, 1971) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The MAST is a 25-item questionnaire which aims to screen for lifetime alcohol-related problems and alcoholism.
Change in Fagerstrom Test for Nicotine Dependence and Heaviness of Smoking (FTQ; Heatherton et al., 1991) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The FTQ provides a brief self-report measure of nicotine dependence.
Change in Yale Food Addiction Scale (YFAS; Gearhardt et al., 2009) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The YFAS purports to assess markers of substance dependence in relation to the consumption of high fat and high sugar foods.
Change in Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The DERS is a 36- item self-report measure of emotion dysregulation, providing a total score and six subscale scores: limited access to adaptive emotion regulation strategies, lack of emotional clarity, lack of emotional awareness, impulse control problems when distressed, problems maintaining goal-focused behavior when distressed, and non-acceptance of negative emotions.
Change in UPPS-P Impulsive Behavior Scale (UPPS-P; Whiteside & Lynam, 2001) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The UPPS-P is a 59-item self-report questionnaire that assesses five different kinds of impulsivity: negative urgency, positive urgency, sensation seeking, lack of perseverance, and lack of premeditation.
Change in Adult Temperament Questionnaire-Short Form (ATQ-SF; Evans & Rothbart, 2007) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The ATQ-SF is a self-report measure of adult temperament traits that contains several subscales. In the current study, only the 19-item Effortful control subscale will be used, which assesses attentional control, control over behavioral activation, and control over behavioral inhibition.
Change in Emotional Eating Scale (EES; Arnow, Kenardy, & Agras, 1995) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The EES is a self-report measure which purports to assess the extent to which individuals cope with negative affect through eating behavior. It includes three subscales: Anger/Frustration, Anxiety, and Depression.
Change in Eating Disorder Examination Overeating Section (EDE; Fairburn, 2008) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The overeating section of the EDE will be used to assess overeating, binge eating, and loss of control eating in this sample.
Change in SCID-I/P Impulse Control Module (First et al., 1995; Muller et al., 2009) | Pre-surgery (up to 3 months before surgery) and 1 year post surgery
  The Impulse Control module will be used to measure compulsive buying, gambling, trichotillomania, skin picking, shoplifting, internet use, sexual behavior, intermittent explosive disorder, kleptomania, and pyromania.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Steffen, PharmD, PhD, Principal Investigator — Neuropsychiatric Research Institute; Scott Engel, PhD, Principal Investigator — Neuropsychiatric Research Institute
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States